CLINICAL TRIAL: NCT06802380
Title: Neuromodulation in Patients With Pulmonary Arterial Hypertension
Acronym: NIP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17677; 17677 (Other: OUHSC IRB)
Record Dates: First submitted 2024-12-06; First posted 2025-01-31 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension
Keywords: Neuromodulation; Endothelial function; 6-minute walk distance; Right ventricular function
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Randomized clinical study using low-level tragus stimulation compared to sham stimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patient's and principal investigator and outcomes assessor will be blinded to the allocation am of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LLTS arm (Experimental): Patients in this group will undergo low-level tragus stimulation for 1 hour every day for 4 weeks.
  Interventions: Device: Low-level tragus stimulation
- Placebo arm (Sham Comparator): Patient will undergo stimulation but on the ear lobule which is devoid of any vagus nerve innervation. This will be used as a sham comparison group.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Low-level tragus stimulation — Low-level tragus stimulation will recruit the fibers from the inner part of the tragus of the external ear and sent afferent signals through the greater auricular branch of the vagus nerve. Ultimately the stimulation is transmitted to the dorsal vagal complex and the brainstem thereby modulating the neuronal activity in the vehicle output. Sham stimulation will be performed by clipping the electrode to the ear lobule which will not relay any afferent signals through the greater auricular branch of the vagus nerve.
  Arms: LLTS arm
Device: Sham stimulation — In the sham stimulation the electrodes will be attached to the ear lobule which are devoid of any afferent nerves traveling to the greater auricular branch of the vagus nerve.
  Arms: Placebo arm

SUMMARY:
Patients with Group 1 pulmonary hypertension will be enrolled in this study. Investigators will test the hypothesis of low-level tragal stimulation in patients with pulmonary hypertension. The study will be conducted over 4 weeks and patients will undergo low-level tragus stimulation for 1 hour every day for 4 weeks. At baseline the following tests will be conducted-6-minute walk distance, vascular function testing using noninvasive device and blood samples will be collected. Patient will also undergo a limited echocardiography to assess right ventricular function. After 4 weeks of stimulation patients will come back to undergo these tests again. Investigators hypothesized that low-level tragus stimulation (neuromodulation) will lead to improvement in vascular function, 6-minute walk distance and blood based biomarkers in patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Investigators propose the following aims:

Aim 1: Quantitatively measure effects of LLTS on exercise capacity and quality of life in Pulmonary hypertension. A 6MWD and QoL (using Pulmonary hypertension questionnaire) will be performed at baseline and follow up (1 months).

Hypothesis 1: Short term LLTS would lead to improvement in exercise capacity and QoL.

Aim 2: Measure effect of neuromodulation on autonomic tone and inflammation. Heart rate variability (frequency and time domains) will be measured at baseline and after 1 months of LLTS. Serum will be used to analyze NT-Pro BNP, circulating inflammatory markers (IL-6,IL-18,TNF-a, IL1ra and CRP).

Hypothesis 2: Short term LLTS would lead to improvement in autonomic tone and inflammation.

Aim 3: Measure the effect of LLTS on endothelial function . Endothelial function (using ENDOPAT test) will be determined at baseline and at 1 months.

Results from this study will help investigators better understand PAH pathogenesis and provide investigators with further therapeutic targets and opportunities.

EXPERIMENTAL DESIGN:

For this application, investigators propose a prospective randomized double-blind study of LLTS vs. sham treatment.

Inclusion criteria: Patients older than 18 years of age, with pulmonary arterial hypertension (Group 1 PH) and WHO functional class II/III Exclusion:Patients with Inability to walk, wheelchair-bound, amputations, expected survival less than 3 to 6 months, active malignancy patients who are Spanish-speaking. would be excluded from the study.

PROPOSED PROCEDURE:

Patients with PAH would be screened from the Pulmonary Hypertension clinic located at OU Physicians building by the pulmonary hypertension facutly. Patients who meet inclusion criteria and consent to the study would be recruited.

Demographic data, medications used for PH, co-morbid conditions would be recorded. Patients would be escorted to the cardiovascular lab at the O-Donoghue building by the PH co-ordinator. EKG for heart rate variability, Six minute walk test, Endopat test for endothelial dysfunction would re recorded. The visit is expected to take close to 60 minutes.

Device administration and treatment protocol: Subjects will be trained on the day of enrollment to use PARASYM unit for self-administration of LLTS. Investigators will spend ample time explaining the nuances of the devices and provide time to subjects to familiarize with the device. Patients will be instructed to apply LLTS to the Tragus or ear lobe. Instruction manual and batteries will be provided.

In case of device malfunction, new devices will be provided to subjects within 48-72 hours (via mail or in person). Device parameters will be set to pulse width of 200 us and pulse frequency of 20 Hz. Amplitude will be titrated to level of sensory threshold (minimum 1 mA). The frequency and pulse width settings have been chosen based on our preliminary studies of LLTS in atrial fibrillation, diastolic HF and systolic HF. The final stimulation strength will be below the threshold (final output ³1mA) and subjects will be barely able to sense it. Patients will maintain a diary log for 4 weeks and perform stimulation for 1 hour daily (typically between 4-8pm, during the 2nd diurnal phase of high sympathetic tone). The time between 4-8 pm was selected for patient convenience as certain patients work hours may restrict use during the first diurnal phase in the morning. Sympathetic tone is highest during these diurnal phases, hence the rationale to target therapy during those times. The PARASYMTM device is also equipped with a treatment time recorder to get accurate logs of treatment. Patients will be asked to avoid caffeine for 4 hrs. and alcohol, smoking, and exercise for 12 h before the visit to avoid any interference with the functional tests that are performed

ELIGIBILITY:
Inclusion criteria: Patients older than 18 years of age, with pulmonary arterial hypertension (Group 1 PH) and WHO functional class II/III

Exclusion:Patients with Inability to walk, wheelchair-bound, amputations, expected survival less than 3 to 6 months, active malignancy patients who are Spanish-speaking. would be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 4 weeks
  Change in the heart rate variability metrics. These are reflective of the autonomic tone and the imbalance. Investigators hypothesized that using low-level tragus stimulation in patients with pulmonary hypertension the heart rate variability will be favorably affected using low-level tragus stimulation compared to sham stimulation.
  Time domain metrics are usually measured using variation of the standard R-R interval on the EKG in milliseconds.

SECONDARY OUTCOMES:
6-minute walk distance | 4 weeks
  A 6-minute walk test will be performed and the distance walked in 6 minutes as measured in meters will be quantified. Investigators hypothesized that using low-level tragus stimulation 6-minute walk distance will improve in patients with pulmonary hypertension after using the device for 4 weeks. This is in comparison to sham stimulation.

OTHER OUTCOMES:
Right ventricular function | 4 weeks
  Using low-level tragus stimulation and pulmonary hypertension for 4 weeks, Investigators hypothesized that L LTS will lead to improvement in right ventricular mechanics and function.This will be assessed using echocardiography and right ventricular function metrics using right ventricular ejection fraction (%) will be assessed.
Endothelial oxidative stress | 4 weeks
  Using low-level tragus stimulation and pulmonary hypertension for 4 weeks, investigators hypothesized that L LTS will lead to improvement in Endothelial oxidative stress. This will be assessed using vascular function assays that measure oxidative stress using units termed MITOSOX. This will be expressed as a continuous numerical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Dasari, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma health sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided